CLINICAL TRIAL: NCT00341419
Title: Genetic Analysis of Patients With Pseudoxanthoma Elasticum (PXE)
Brief Title: Genetic Analysis of Patients With Pseudoxanthoma Elasticum
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905106; 05-C-N106
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-05-14

CONDITIONS: Pseudoxanthoma Elasticum; PXE
Keywords: ABC Transporter; ABCC6; Slkin Laxity; Genetic Association; Angiod Streaks; Pseudoxanthoma Elasticum; PXE
MeSH Terms: conditions — Pseudoxanthoma Elasticum

SUMMARY:
This study will characterize the gene mutations responsible for pseudoxanthoma elasticum (PXE) and correlate them with disease manifestations in males and females. PXE is an inherited disorder that affects the connective tissue in some parts of the body. Calcium and other minerals are deposited in the connective tissue, causing changes in the skin, eyes, cardiovascular system and gastrointestinal system. Some effects of PXE can cause serious medical problems, while others have less impact. Symptoms often appear earlier and are more severe in females than in males, but there is no way to predict how the disorder will progress in any given individual.

Candidates for this study are recruited through PXE International, an organization that provides patient support and supports research on the disease. The organization collects biological samples and medical information on patients and family members to help further research on the disease. Families that have samples from the patient, both parents, and at least one sibling may be eligible for this study. Grandparents and extended family members may be included in certain instances.

Participants provide a blood sample, a sample of cells scraped from the inside of the cheek (buccal cells) and a medical history. The samples are analyzed for gene variants and the findings are correlated with disease signs and symptoms.

...

DETAILED DESCRIPTION:
Background:

* Pseudoxanthoma elasticum (PXE) is an autosomal recessive genetic disorder characterized by mutations in the ATP-binding cassette transporter, ABCC6.
* PXE while it is known that patients have two mutated alleles of the ABCC6 gene, significant questions remain about the segregation of the disease, the presentation in males versus females and the correlation of mutation to clinical phenotype.

Objectives:

- The objective is to examine the role of variants in the ABCC6 gene in PXE.

Eligibility:

* Samples from study participants were obtained through the PXE International BioBank.
* Families were selected that have samples from both parents and at least one sibling in addition to the proband.

Design:

- Participants DNA was sequenced to identify variants and genotyped for linked markers to follow the segregation of mutant alleles and compare the results with the clinical outcomes.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

A representative set of collected families will be studied. No subjects within these families will be excluded.

Families will be selected that have samples from both parents and at least one sibling in addition to the proband.

The siblings will include both affected and unaffected.

If grandparents are available they will also be typed to help in phase determination.

Extended relatives will only be selected in multiple generation families.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2005-02-16; Study Completion 2013-05-14

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dean, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hagedorn C. Influences of soil acidity on Streptomyces populations inhabiting forest soils. Appl Environ Microbiol. 1976 Sep;32(3):368-75. doi: 10.1128/aem.32.3.368-375.1976. PMID 10835
- [Background] Dean M, Rzhetsky A, Allikmets R. The human ATP-binding cassette (ABC) transporter superfamily. Genome Res. 2001 Jul;11(7):1156-66. doi: 10.1101/gr.184901. PMID 11435397
- [Background] Bodzioch M, Orso E, Klucken J, Langmann T, Bottcher A, Diederich W, Drobnik W, Barlage S, Buchler C, Porsch-Ozcurumez M, Kaminski WE, Hahmann HW, Oette K, Rothe G, Aslanidis C, Lackner KJ, Schmitz G. The gene encoding ATP-binding cassette transporter 1 is mutated in Tangier disease. Nat Genet. 1999 Aug;22(4):347-51. doi: 10.1038/11914. PMID 10431237